CLINICAL TRIAL: NCT06093360
Title: Flapless Surgical Approach in the Treatment of Peri-implantitis
Brief Title: Flapless Surgical Treatment of Peri-implantitis
Status: Completed | Type: Observational
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Ana Carrillo de Albornoz, Flapless surgical approach in the treatment of peri-implantitis., Universidad Complutense de Madrid
Other Study IDs: UCM ACA 2
Record Dates: First submitted 2023-10-09; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Peri-Implantitis
Keywords: treatment; systemic antimicrobials
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- flapless group: Patients were treated in 1-2 sessions within a period of 7 days, with a minimum of 90 minutes per session. Implant-supported restorations were unscrewed and modified if they were not cleansable. After local anesthesia, a periodontal ultrasonic stainless-steel tip was used for supra- and sub-mucosal mechanical debridement . Next, a Columbia 4R/4L curette was used around the implant in a circular motion until a bone exposure of 2-3 mm was achieved. Mucosal curettage was performed. After obtaining access to the implant surface, ultrasonic instrumentation was repeated and air polishing with an erythritol powder was applied submucosally with the aim of a periodontal probe. Hydrogen peroxide 3% was used to irrigate the implant surface for 2 minutes, followed by a rinse with saline. Systemic antibiotics, when prescribed, were metronidazole or azithromycin.
  Interventions: Procedure: flapless surgery

INTERVENTIONS:
Procedure: flapless surgery — Implant-supported restorations were unscrewed and modified if necessary (biofilm control). All the restorations were relocated at the end of each intervention session. After local anesthesia, a periodontal ultrasonic stainless-steel tip was used for supra- and sub-mucosal mechanical debridement. Next, a Columbia 4R/4L curette was used around the implant in a circular motion until a bone exposure of 2-3 mm was achieved. Mucosal curettage was simultaneously performed to remove the granulation tissue. After obtaining access to the implant surface, ultrasonic instrumentation was repeated and air polishing with an erythritol powder was applied submucosally with the aim of a periodontal probe. Hydrogen peroxide 3% was used to irrigate the implant surface for 2 minutes, followed by a rinse with saline. Oral hygiene instructions were given. Systemic antibiotics, when prescribed, were metronidazole or azithromycin

SUMMARY:
Aim: To evaluate the effectiveness of a flapless surgical approach in the treatment of peri-implantitis and to explore the factors influencing disease resolution.

Material and Methods: This case series involved patients with at least one implant diagnosed with peri-implantitis treated with a flapless surgical approach. Treatment consisted on mechanical debridement and chemical decontamination of the implant surface plus mucosal curettage combined with/without systemic antimicrobials and/or prostheses modification. Follow-up visits for supportive peri-implant care (SPIC) were scheduled at 6 and 12 weeks, and then every 3 months during the first 12 months. Clinical and radiographic parameters were assessed at baseline, 3 months and 12 months. Disease resolution defined as residual probing depths < 5 mm, ≤ 1 point of BOP, absence of suppuration and absence of progressive bone loss compared to pre-treatment bone levels was the main outcome variable. Multilevel regression analyses was used to identify predictors affecting the probability of disease resolution.

DETAILED DESCRIPTION:
INTRODUCTION

Peri-implant diseases, especially peri-implantitis, represent a growing public health problem due to their high prevalence and the associated consequences (implant and implant-supported prosthesis loss). In addition, given the complex histopathology and the accelerated pattern of disease progression, peri-implantitis is considered one of the most challenging biological complications to treat.

A step-by-step approach has been proposed in the Clinical Practice Guidelines to maintain healthy peri-implant tissues and to manage peri-implant diseases, recommending that the treatment of peri-implantitis should start with a non-surgical step. However, systematic reviews have shown limited predictability and conflicting results for non-surgical treatment , suggesting that clinical and patient-reported benefits remain to be proven. Consequently, surgical interventions are frequently recommended due to the advantage of gaining access to remove the biofilm from the implant surface. However, treatment success based on clinical and radiographic outcomes,, for patients enrolled in regular post-treatment supportive care, are within 33-75% at the implant level following non-reconstructive surgical protocols and 51-58% with surgical reconstructive therapy.

To compensate the limited access to the implant surface, recent studies are including the curettage as part of the non-surgical treatment with promising results. With this procedure the granulation tissue is removed from the peri-implant mucosa and, if extended, it can also detach the periosteum and obtain direct access to the crestal bone and the entire contaminated implant surface. Given the inability of the peri-implant connective tissue to separate the inflammatory cell infiltrate from the crestal bone, gaining access to this critical area with a low morbidity procedure may represent an interesting alternative treatment strategy. With this modification, the treatment may be considered a minimally invasive surgery, with clear advantages for the patient in comparison to conventional open flap surgical techniques. This treatment strategy, however, needs to be further studied.

The objective of this case series was to evaluate the effectiveness of a flapless surgical approach in patients with peri-implantitis in terms of disease resolution and to explore the involved factors after a follow-up of 12 months.

MATERIAL AND METHODS

Study design and ethical considerations

This retrospective case-series was reported according to the Strengthening the Reporting of Observational studies in Epidemiology guidelines and was conducted in accordance with the Declaration of Helsinki. Written informed consent was obtained in accordance with local standards, along with local ethical committee approval

Patient screening

Patients referred to a private practice in Madrid, Spain, for the treatment of peri-implantitis and who met the inclusion criteria were consecutively recruited from from January to June 2023, were recruited for the study. The inclusion criteria for patients were as follows: i) > 18 years old; ii) presence before treatment of at least one implant diagnosed with peri-implantitis following the case definition of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions, defined as probing pocket depth > 6 mm combined with bleeding on probing and/or suppuration and progressive bone loss in relation to the radiographic bone level assessment at 1 year following the delivery of the implant-supported prosthetics reconstruction. In the absence of initial radiographs, radiographic evidence of bone level ≥3 mm was considered; iii) follow-up period after treatment of at least 12 months. Subjects were excluded if they were i) pregnant or breast-feeding; ii) had systemic contraindications to receive treatment; iii) had presence of implant-supported removable overdentures; iv) present implant mobility before treatment; or v) present inability or unwillingness to give informed consent.

Intervention

A single experienced periodontist with 2.5 X magnification loops performed the interventions in all the patients. Patients were treated in 1-2 sessions within a period of 7 days, with a minimum of 90 minutes per session. Implant-supported restorations were unscrewed when full access to the implant surface and surrounding bone crest was not guaranteed. Unscrewed prostheses were modified in the laboratory if they were not cleansable (allowing implant hygiene access for biofilm removal) or to eliminate/reduce porcelain in direct contact with the bone when it was present. All the restorations were relocated at the end of each intervention session. After local anesthesia, a periodontal ultrasonic stainless-steel tip was used for supra- and sub-mucosal mechanical debridement . Next, a Columbia 4R/4L curette was used around the implant in a circular motion until a bone exposure of 2-3 mm was achieved. Mucosal curettage was simultaneously performed to remove the granulation tissue adjacent to the contaminated implant surfaces. After obtaining access to the implant surface, ultrasonic instrumentation was repeated and air polishing with an erythritol powder was applied submucosally with the aim of a periodontal probe to separate and retract the peri-implant mucosa during the procedure. Hydrogen peroxide 3% was used to irrigate the implant surface for 2 minutes, followed by a rinse with saline. Oral hygiene instructions were given in detail at the end of the treatment. Systemic antibiotics, when prescribed, were metronidazole 500 mg every 8 h for 7 days or azithromycin 500 mg every 24 h for 3 days. If patients were already taking amoxicillin or need antibiotic prophylaxis for systemic reasons, it was maintained until the prescription ended (7 days).

Supported peri-implant care program

Follow-up visits for SPIC were scheduled at 6 and 12 weeks, and then every 3 months during the first 12 months. After 12 months and according to the patient risk profile, SPIC was recommended every 3-6 months. Oral hygiene was individually reinforced at each visit as needed.

Sites with residual PPD > 5 mm with BOP after 3 months were re-instrumented as previously described without any further systemic antibiotic. Implants presenting progressive clinical and/or radiographic worsening despite re-instrumentation were referred for an open flap debridement procedure or for explantation in case implants were mobile or broken during the follow-up (including those adjacent implants becoming useless due to restorable reasons).

Data collection

Baseline patient and implants characteristics

At baseline, the following patient characteristics were registered: age, gender, smoking habit, number of cigarettes per day, presence/absence of potentially related systemic diseases (i.e. diabetes, hypothyroidism, osteoporosis, anxiety and/or depression disorders), diagnosis of periodontitis, periodontitis stage (I-IV), if the patient was periodontally stable defined as bleeding on probing < 10% of sites, no probing depths > 4 mm that bleed on probing and lack of progressive periodontal destruction, type of toothbrush (manual or powered) and full mouth plaque score.

The following characteristics of the included implants were recorded at baseline: implant site (anterior, premolar, molar), implant arch (maxilla, mandible), implant diameter (i.e < 4 mm, > 4 and < 5mm or > 5 mm), type of prosthesis (single crown, fixed partial prosthesis), prosthesis retention (screw retained/cemented), time since implant placement, prosthesis material (i.e. metal-porcelain, zirconia or metal-resin), access to oral hygiene before treatment, prosthesis removal during the treatment, prosthesis modification as part of the treatment, vestibule depth (i.e. shallow or deep), presence of keratinized mucosa (< 2 mm or > 2 mm), presence of intermediate abutment and abutment height (< 2 mm or > 2 mm).

Clinical parameters

A previously calibrated examiner carried out all clinical measurements. Patients were examined for peri-implant parameters pre-operatively and twice post intervention, at 3 months and 12 months after treatment. Implants were measured using a UNC 15 manual periodontal probe at six sites per implant to the nearest mm for probing pocket depth and dichotomously scored at six sites per implant for bleeding on probing , suppuration and presence/absence of biofilm detected by the periodontal probe (implant plaque score).

Radiographic parameters

Measurements of radiographic outcomes were done by an independent and calibrated examiners. The calibration exercise consisted on repeated measurements of 40 randomly selected radiographs. The achieved inter-examiner intraclass correlation coefficient for marginal bone levels was 0.99 (95% confidence interval: [0.97; 0.99]). Standardized intra-oral periapical radiographs were taken using a long-cone paralleling technique. The radiographs were taken before intervention and at 12 months after treatment. Each radiograph was calibrated using the implant length as the fixed reference and the following linear measurements were carried out using an image analysis software to the nearest 0.1 mm: i) marginal bone levels (vertical distance expressed in mm from the implant shoulder to the most coronal interproximal bone implant contact at mesial and distal sides); ii) vertical intra-bony defect depth (vertical linear distance expressed in mm measured from the bone crest to the most coronal interproximal bone implant contact at mesial and distal sides); and iii) intra-bony defect width (horizontal linear distance expressed in mm measured between the mesial and distal interproximal bone crest and the implant surface).

Disease resolution

The endpoint of the treatment and primary outcome of the study was the composite outcome disease resolution, defined as concomitant residual probing depths < 5 mm, < 1 point of BOP, absence of suppuration and absence of progressive bone loss compared to pre-treatment bone levels.

Data Analyses

Clinical and radiographic parameters were expressed as means and standard deviations for continuous variables and as absolute and relative frequencies for categorical variables at baseline, 3-months and > 12 months. Differences were analyzed using analysis of variance and the chi-squared test. Adjustment for multiple comparisons (pairwise tests) were performed using the Bonferroni correction method. A p value <0.05 was considered as statistically significant.

The primary outcome variable was disease resolution at the last follow-up examination. To identify factors affecting the probability of treatment success, a multiple logistic multilevel model was used. The hierarchical analysis included the patient at the higher level and the implant at the lower level. The logit function was applied to link the linear model with the probability of the binary event. The independent factors examined included treatment factors (i.e. systemic antimicrobial prescribed), patient-related data (age, gender, smoking habit, systemic diseases, diagnosis of periodontitis, use of manual or powered-toothbrushes, full-mouth plaque score and compliance with supportive peri-implant care program), and implant- and prostheses-related data (number of affected implants, jaw, location, implant surface and diameter, time since implant placement, type of prostheses, prostheses retention and material, etc.). The model was built with the intercept as a random term. All variables were assessed by the Wald test in a bivariate analysis, and only statistically significant variables (P < 0.05) were retained in the multiple model. The treatment factor (i.e the systemic antimicrobial prescribed, if any) were forced into the final model, and a possible interaction between the factor and the covariates was explored. Results were expressed as odds ratios (ORs) including 95% confidence intervals (CIs).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* presence before treatment of at least one implant diagnosed with peri-implantitis following the case definition of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions, defined as probing pocket depth > 6 mm combined with bleeding on probing and/or suppuration and progressive bone loss in relation to the radiographic bone level assessment at 1 year following the delivery of the implant-supported prosthetics reconstruction. In the absence of initial radiographs, radiographic evidence of bone level ≥3 mm was considered; - follow-up period after treatment of at least 12 months

Exclusion Criteria:

* pregnant or breast-feeding
* had systemic contraindications to receive treatment
* had presence of implant-supported removable overdentures
* present implant mobility before treatment
* present inability or unwillingness to give informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with peri-implantitis in need of treatment
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Disease resolution percentage | 12 months, 60 months
  Percentage of implants that achieve disease resolution, defined as:probing depths < 5 mm + < 1 point of bleeding on probing (BOP) + absence of suppuration and absence of progressive bone loss compared to pre-treatment bone levels

SECONDARY OUTCOMES:
Probing deph | baseline, 3 months, 12 months, 60 months
  Measurement with a periodontal probe the distance: soft tissue margin to the bottom of the sulcus
bleeding on probing | baseline, 3 months, 12 months, 60 months
  Measurement of bleeding after probing, at six sites per implant
recession | baseline, 3 months, 12 months, 60 months
  measurement with a periodontal probe of the distance from implant shoulder to the mucosal soft tissue margin
suppuration | baseline, 3 months, 12 months, 60 months
  Measurement of suppuration after probing, at six sites per implant
marginal bone levels | Baseline, 12 months
  vertical distance expressed in mm from the implant shoulder to the most coronal interproximal bone implant contact at mesial and distal sides (measured in periapical X-ray)
vertical intra-bony defect depth | Baseline, 12 months
  vertical linear distance expressed in mm measured from the bone crest to the most coronal interproximal bone implant contact at mesial and distal sides, measured in standardized periapical X-Ray
intra-bony defect width | Baseline, 12 months
  horizontal linear distance expressed in mm measured between the mesial and distal interproximal bone crest and the implant surface, measured in periapical X-ray
Age | Baseline
  Age of the patients
Gender | Baseline
  Male/female
smoking habit | Baseline
  yes/no/number of cigarettes per day
potentially related systemic diseases | Baseline
  Yes/no
diagnosis of periodontitis | Baseline
  Yes/no
stage of periodontitis | Baseline
  I, II, III, IV
periodontally stable patient | Baseline
  Yes/no defined as bleeding on probing < 10% of sites, no probing depths > 4 mm that bleed on probing and lack of progressive periodontal destruction)
Type of toothbrush | Baseline
  electronic, manual
Bull mouth of plaque score | Baseline
  Presence /absence of dental biofilm (percentage)
Implant site | Baseline
  Anterior, premolar, molar
Implant arch | Baseline
  Maxilla/mandible
Implant diameter | Baseline
  < 4 mm, > 4 and < 5mm or > 5 mm
Type of prosthesis | Baseline
  single crown, fixed partial prosthesis
Prosthesis retention | Baseline
  screw retained/cemented
time since implant placement | Baseline
  Number of years after implants were placed
prosthesis material | Baseline
  metal-porcelain, zirconia or metal-resin)
access to oral hygiene before treatment | Baseline
  Yes/no
prosthesis removal during the treatment | Baseline
  Yes/no
prosthesis modification as part of the treatment | Baseline
  Yes/no
prosthesis modification as part of the treatment | Baseline
  prosthesis modification as part of the treatment
presence of keratinized mucosa | Baseline
  < 2 mm or > 2 mm
presence of intermediate abutment | Baseline
  Yes/no
Abutment height | Baseline
  < 2 mm, > 2 mm

CONTACTS AND LOCATIONS:
Locations (1):
- Ana Carrillo de Albornoz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Share of the protocol, results will be available in the publication

REFERENCES:
- [Result] Herrera D, Berglundh T, Schwarz F, Chapple I, Jepsen S, Sculean A, Kebschull M, Papapanou PN, Tonetti MS, Sanz M; EFP workshop participants and methodological consultant. Prevention and treatment of peri-implant diseases-The EFP S3 level clinical practice guideline. J Clin Periodontol. 2023 Jun;50 Suppl 26:4-76. doi: 10.1111/jcpe.13823. Epub 2023 Jun 4. PMID 37271498